CLINICAL TRIAL: NCT06574360
Title: Dual Modulation of Sigma-1 and NMDA Receptors in the Treatment of Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH112-REC3-202
Record Dates: First submitted 2024-08-25; First posted 2024-08-27 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; sigma-1 receptor
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1R agonist (S1RA) plus NMDAE (Experimental): An S1R agonist plus an NMDA enhancer
  Interventions: Drug: S1RA plus NMDAE
- S1R agonist (S1RA) plus placebo (Placebo Comparator): An S1R agonist plus placebo
  Interventions: Drug: S1RA plus Placebo Cap

INTERVENTIONS:
Drug: S1RA plus NMDAE — Use of an S1R agonist plus an NMDA enhancer for the treatment of treatment-resistant schizophrenia.
  Arms: S1R agonist (S1RA) plus NMDAE
Drug: S1RA plus Placebo Cap — Use of an S1R agonist plus placebo as a comparator
  Arms: S1R agonist (S1RA) plus placebo

SUMMARY:
sigma-1 receptor (S1R) agonistic property have been tested in clinical trials for the treatment of schizophrenia. In addition, previous studies found that some NMDA receptor (NMDAR)-enhancing agents were able to improve clinical symptoms of patients with chronic schizophrenia. Whether combined treatment of an S1R agonist and an NMDA-enhancing agent can be better than an S1R agonist alone deserves study.

DETAILED DESCRIPTION:
The current treatment for schizophrenia remains unsatisfactory; thus, development of new treatments is vital. Both sigma-1 receptor (S1R) dysfunction and NMDA receptor (NMDAR) hypofunction contribute to pathogenesis of schizophrenia, especially treatment-resistant schizophrenia. Several S1R agonists have been tested for its potential for schizophrenia treatment; however, its efficacy appears limited. In addition, previous studies also found that some NMDA-enhancing agents were able to augment efficacy of antipsychotics in the treatment of chronic schizophrenia. Whether combined treatment of an S1R agonist and an NMDA-enhancer (NMDAE) can be better than an S1R agonist alone deserves study. Therefore, this study aims to compare an S1R agonist plus an NMDAE and an S1R agonist plus placebo in the treatment of treatment-resistant schizophrenia. The subjects are the patients with treatment-resistant schizophrenia who have responded poorly to two or more kinds of antipsychotics treatment. They keep their original treatment and are randomly, double-blindly assigned into two treatment groups for 12 weeks: (1) S1R agonist (S1RA) plus NMDAE, or (2) S1RA plus placebo. Clinical performances and side effects are measured at weeks 0, 2, 4, 6, and 8. Cognitive functions are assessed at baseline and at endpoint of treatment by a battery of tests. The efficacies of S1RA plus NMDAE and S1RA plus placebo will be compared.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a DSM-5 (American Psychiatric Association) diagnosis of schizophrenia
* Are resistant to adequate treatments of at least two antipsychotics (excluding clozapine)
* Remain symptomatic but without clinically significant fluctuation, while their antipsychotic doses are unchanged for at least 3 months and will be maintained during the period of the 8-week trial
* PANSS total score >70
* Hamilton Depression Rating Scale-17 items (HAMD) <7
* Are physically healthy and laboratory assessments (including blood routine, biochemical tests) are clinically insignificant.
* Have sufficient education to communicate effectively and are capable of completing the assessments of the study.
* Agree to participate in the study and provide informed consent

Exclusion Criteria:

* DSM-5 diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, central nervous system diseases or mental disorders other than schizophrenia (including major depressive disorder, bipolar disorders, persistent depressive disorder, obsessive-compulsive disorder)
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 2, 4, 6, 8
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change of scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 2, 4, 6, 8
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Positive subscale, Negative subscales, and General Psychopathology subscale of PANSS | week 0, 2, 4, 6, 8
  PANSS-positive: Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-negative: Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
  PANSS-general psychopathology: Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome.
Clinical Global Impression | week 0, 2, 4, 6, 8
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Global Assessment of Functioning | week 0, 2, 4, 6, 8
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Quality of Life Scale | week 0, 2, 4, 6, 8
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.
Cognitive function | Week 0, 8
  Ten tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, Wechsler Adult Intelligence Scale(WAIS)-III Digit Symbol-Coding)
  2. sustained attention (Continuous Performance Test)
  3. working memory: verbal (digit span) and nonverbal (spatial span)
  4. verbal learning and memory (WMS-III, word listing)
  5. visual learning and memory (WMS-III, visual reproduction)
  6. reasoning and problem solving (WISC-III, Maze)
  7. social cognition (MSCEIT Version 2)
  For the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score. Furthermore, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains) will be also calculated by standardizing the average of the T score (Lane HY et al, JAMA Psychiatry 2013)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan